CLINICAL TRIAL: NCT06590779
Title: Evaluation of the Benefits of a Cosmetic Anti-hair Loss Lotion Applied in Combination With Finasteride in Male Subjects With Hair Loss: Investigator-blinded, Randomized, Multi-center Study Performed Under Dermatological Control
Brief Title: Benefits of a Cosmetic Anti-hair Loss in Males With Hair Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCY23-015
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Finasteride

STUDY DESIGN:
Intervention Model Description: Arm 1: Finasteride 1mg Arm 2: Finasteride 1mg + Aminexil® active+ lotion
Who Masked: Investigator
Masking Description: Investigator blinded, randomised study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finasteride 1 mg & Aminexil® active+ lotion (Experimental): Administration of Finasteride 1 mg + Aminexil® active+ lotion
  Interventions: Other: Aminexil® active+ lotion; Other: Finasteride 1mg
- Finasteride 1 mg (Active Comparator): Administration of Finasteride 1 mg
  Interventions: Other: Finasteride 1mg

INTERVENTIONS:
Other: Aminexil® active+ lotion — Aminexil® active+ lotion
  Arms: Finasteride 1 mg & Aminexil® active+ lotion
Other: Finasteride 1mg — Finasteride 1 mg

SUMMARY:
Androgenetic alopecia (AGA), also known as androgenic alopecia or male pattern baldness, is the most common type of progressive hair loss. AGA is a polygenetic condition with varying severity, age of onset, and scalp location of hair loss. In men, hair loss typically involves the temporal and vertex region while sparing the occipital region: the characteristic "horseshoe" pattern. Incidence and prevalence of AGA depend on age and race.

Vichy has developed a new cosmetic anti hair loss lotion with the aim of acting on androgenic alopecia. The aim is to improve the efficacy on hair loss of the association of the lotion with finasteride versus finasteride alone.

The primary objective of this investigator-blinded, randomized multi-center study is to quantitatively evaluate, using the phototrichogram method, the efficacy of a lotion associated with finasteride versus finasteride alone on hair growth parameters in male subjects with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged 18-41 years old with skin type I to IV according to the Fitzpatrick scale;
* Affected by androgenetic alopecia with hair loss evaluated grade IIA to IV the modified Norwood-Hamilton scale;
* Subject with chestnut brown, dark or black hair;
* Subject with hair length ≥ 3 cm on the vertex and agreeing to keep this minimum length for the duration of the study;
* Subject agreeing to have a shaved zone of 1.5 cm² on scalp area;
* Subject accepting not to dye, bleach his hair or to do a permanent wave during the whole study duration;
* Subject accepting to use condoms if her partner is pregnant.

Exclusion Criteria:

* Female subject;
* Subject presenting a life-threatening endocrine disease, neoplasia or other serious diseases;
* Subjects suffering from chemo-induced alopecia (poisoning, medicines), or resulting from a chronic disease (genetic, endocrine, immunological, deficiencies), seasonal hair loss;
* Subject having any other concomitant dermatological affection of the scalp (psoriasis, seborrheic dermatitis, eczema, other alopecia than androgenetic);
* Subject suffering from a recurrent, acute, non-stabilized or evolving disease judged by the investigator able to interfere with the study needs and hair growth;
* Subject having had surgical intervention for capillary correction (e.g., hair transplant) or intending to have recourse to this surgery during the entire study period;
* Subject presenting a hypersensitivity to any of the components of the finasteride medication or to any 5-alpha-reductase inhibitor;
* Subject that has applied or taken prior to the start of the study (screening) interfering drugs or products
* Subject taking any other medical treatment (topic or per os) likely to interfere on hair growth or hair loss within 6 months prior to the screening visit;
* Subject following a long period (>30 days) treatment of anti-inflammatory within 4 months prior to the start of the study (screening visit);
* Subject taking topic cosmetic treatment or per os nutritional supplement likely to interfere on hair growth or hair loss during the last 3 months prior to the screening visit;
* Subject having a topical or oral route treatment of the scalp (anti-seborrheic, anti-dandruff, daily friction) within 2 weeks prior to the screening visit;
* Subject who has been exposed within one month prior to the screening visit in an intense or excessive manner to sun (natural or artificial) or during the study;
* Subject having a wig or hair extension;
* Protected subject as defined in the Articles of the French Public Health Code. Article 1121-7: person deprived of liberty by a judicial or administrative decision, or subject to psychiatric care, or person admitted to a health or social institution for purposes other than the research. Article 1121-8: adult person subject to a legal protection measure or unable to express his/her consent;
* Subject unable to communicate or cooperate with the Investigator due to poor mental development, language problems or impaired cerebral function;
* Subject currently participating in another clinical study or being in an exclusion period of another clinical study;

Ages: 18 Years to 41 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-02 (Estimated); Primary Completion 2025-12-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Phototrichogram | baseline T0
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 3
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 84
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 86
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 168
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 170
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 336
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles
Phototrichogram | Day 338
  photo of the scalp to assess the rate of hair growth, size of hair fibers and frequency of telogen hair follicles

SECONDARY OUTCOMES:
Scalp coverage evaluation | baseline Day 1
  on a scale 6-point clinical scale from 0: Scalp no visible/Hair completely recovering the scalp to 5:Scalp totally visible
Scalp coverage evaluation | Day 84
  on a scale 6-point clinical scale from 0: Scalp no visible/Hair completely recovering the scalp to 5:Scalp totally visible
Scalp coverage evaluation | Day 168
  on a scale 6-point clinical scale from 0: Scalp no visible/Hair completely recovering the scalp to 5:Scalp totally visible
Scalp coverage evaluation | Day 336
  on a scale 6-point clinical scale from 0: Scalp no visible/Hair completely recovering the scalp to 5:Scalp totally visible
Subject Evaluation on Vertex and Frontal Area of hair quality | baseline Day 1
  scale from -3: greatly decreased to 3: greatly increased
Subject Evaluation on Vertex and Frontal Area of hair quality | Day 84
  scale from -3: greatly decreased to 3: greatly increased
Subject Evaluation on Vertex and Frontal Area of hair quality | Day 168
  scale from -3: greatly decreased to 3: greatly increased
Subject Evaluation on Vertex and Frontal Area of hair quality | Day 252
  scale from -3: greatly decreased to 3: greatly increased
Subject Evaluation on Vertex and Frontal Area of hair quality | Day 336
  scale from -3: greatly decreased to 3: greatly increased
Quality of life assessment | baseline Day 1
  Non-validated 13-point questionnaire; point 1-6: on a 5 point scale from never to always point 7-13 on a 5-point scale from totally agree to not agree at all
Quality of life assessment | Day 84
  Non-validated 13-point questionnaire; point 1-6: on a 5 point scale from never to always point 7-13 on a 5-point scale from totally agree to not agree at all
Quality of life assessment | Day 168
  Non-validated 13-point questionnaire; point 1-6: on a 5 point scale from never to always point 7-13 on a 5-point scale from totally agree to not agree at all
Quality of life assessment | Day 336
  Non-validated 13-point questionnaire; point 1-6: on a 5 point scale from never to always point 7-13 on a 5-point scale from totally agree to not agree at all
Local discomfort | baseline Day 1
  scale from 0: none to 9: hugely
Local discomfort | Day 84
  scale from 0: none to 9: hugely
Local discomfort | Day 168
  scale from 0: none to 9: hugely
Local discomfort | Day 336
  scale from 0: none to 9: hugely
Local reactions | baseline Day 1
  scale from 0: none to 4: very severe
Local reactions | Day 84
  scale from 0: none to 4: very severe
Local reactions | Day 168
  scale from 0: none to 4: very severe
Local reactions | Day 336
  scale from 0: none to 4: very severe
Adverse events | baseline Day 1
  Questioning
Adverse events | baseline Day 3
  Questioning
Adverse events | Day 42
  Questioning
Adverse events | Day 84
  Questioning
Adverse events | Day 86
  Questioning
Adverse events | Day 126
  Questioning
Adverse events | Day 168
  Questioning
Adverse events | Day 170
  Questioning
Adverse events | Day 210
  Questioning
Adverse events | Day 252
  Questioning
Adverse events | Day 294
  Questioning
Adverse events | Day 336
  Questioning
Adverse events | Day 338
  Questioning

IPD SHARING:
Plan to Share IPD: No